CLINICAL TRIAL: NCT01056939
Title: Neurally Adjusted Ventilatory Assist (NAVA) in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Merja Ålander, MD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EETTMK:118/2008
Record Dates: First submitted 2010-01-19; First posted 2010-01-26 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Ventilation
Keywords: Ventilatory care, children, intensive care, NAVA; Children needing ventilatory care
MeSH Terms: conditions — Respiratory Aspiration | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAVA (Active Comparator): Children randomised in this arm will be treated with neurally adjusted ventilatory assist
  Interventions: Device: Neurally adjusted ventilatory assist, i-Servo, Maquet Nordic (Solna, Sweden)
- Control (Active Comparator): Patients randomized to control group will be treated with pressure controlled ventilation (PC) when they are newborns and older children in this group will be treated with pressure regulated volume controlled (PRVC) ventilation.
  Interventions: Device: Control (PC- or PRVC- ventilation), i-Servo, Maquet Nordic (Solna, Sweden)

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist, i-Servo, Maquet Nordic (Solna, Sweden) — Treatment with neurally adjusted ventilatory assist
  Arms: NAVA
Device: Control (PC- or PRVC- ventilation), i-Servo, Maquet Nordic (Solna, Sweden) — Treatment with PC or PRVC ventilation.
  Arms: Control

SUMMARY:
The purpose of this study is to find out if NAVA-technology is better in detecting patients own inspiratory efforts during mechanical ventilation than currently used flow-triggering in PRVC (pressure regulated volume controlled) ventilation, and if NAVA gives real benefits for patients or not.

The investigators study hypothesis is that NAVA-technology can detect spontaneous inspiration more accurately than currently used methods, and thus will lead to more smooth adaptation to mechanical ventilation in pediatric patients. The investigators expect this to decrease the time of ventilatory support needed.

DETAILED DESCRIPTION:
Asynchrony means that the timing of support given by ventilator is different from patients own breathing pattern. Asynchrony during ventilatory care may increase the risk for complications, make the weaning more difficult and may affect the survival rates.

In our study we randomly treat pediatric patients needing ventilatory support with neurally adjusted ventilatory assist and pressure controlled or PRVC-ventilation. We are willing to find out if there are any special benefits for patients with each treatment mode.

ELIGIBILITY:
Inclusion Criteria:

* All children from term newborn (37+0 gestational week) to 16-year-old needing ventilatory care at least 30 minutes

Exclusion Criteria:

* Any condition that prevents feeding tube positioning. Critical ventilatory or perfusion problems.

Ages: 1 Minute to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the duration of mechanical ventilation | 30minutes-3weeks

SECONDARY OUTCOMES:
Amount of sedative medication needed | 30minutes-3weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Oulu, Oulu, Finland